CLINICAL TRIAL: NCT00243945
Title: A Phase 3b, Open-Label, Multicenter, Multinational Trial to Evaluate the Effects of Rotigotine Transdermal Patch on Early Morning Motor Impairment and Sleep Disorders in Patients With Idiopathic Parkinson's Disease
Brief Title: A Trial to Evaluate the Effects of Rotigotine Transdermal Patch on Early Morning Motor Impairment and Sleep Disorders Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0826; 2004-002598-21 (EudraCT Number)
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2009-09

CONDITIONS: IDIOPATHIC PARKINSON'S DISEASE
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

INTERVENTIONS:
Drug: Rotigotine

SUMMARY:
The objective of this trial is to assess the effect of rotigotine (SPM 962) on the control of early morning motor impairment and sleep disorders in subjects with idiopathic PD.

Subjects who meet eligibility criteria will begin treatment with rotigotine transdermal patches. Trial medication will be titrated to an optimal daily dose, or to the maximal dose. Following a Titration period of up to 8 weeks, subjects will be maintained on the optimal or maximal dose for 4 weeks. After the Maintenance period, subjects will have the option to enter into an open-label extension study.

The first subject was enrolled in December 2004. The last subject was enrolled in April 2005 and the last subject visit was conducted in July 2005. This study is now closed

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease

Exclusion Criteria:

* Subject has previously participated in a trial with rotigotine.
* Subject has participated in another trial of an investigational drug within the last 28 days or is currently participating in another trial of an investigational drug.
* Subject discontinued from previous therapy with a dopamine agonist after an adequate length of treatment at an adequate dose due to lack of efficacy as assessed by the investigator.
* Subject has had prior therapy with a dopamine agonist within 28 days prior to Baseline.
* Subject is receiving therapy with controlled-release levodopa within 28 days prior to baseline or is receiving therapy with tolcapone.
* Subject is receiving therapy with one of the following drugs either concurrently or within 28 days prior to Visit 2: alpha-methyl dopa, metoclopramide, reserpine, neuroleptics (including atypical), monoamine oxidase A (MAO-A) inhibitors, methylphenidate, or amphetamine.
* Subject has a history of symptomatic (not asymptomatic) orthostatic hypotension in the 6 months prior to baseline.
* Subject has atypical Parkinsonian syndromes (including drug-induced Parkinsonian syndromes).
* Subject has a history of atopic eczema and/or active skin disease, such as atopic eczema.
* Presence of dementia, active psychosis, or hallucinations (not due to antiparkinsonian medication).
* Subject is receiving CNS therapy (eg, sedatives, hypnotics, selective serotonin reuptake inhibitors [SSRIs], anxiolytics, other sleep-modifying medication) unless dose has been stable daily for at least 28 days prior to baseline and is likely to remain stable for the duration of the trial.
* Subject has a history of seizures or stroke within 1 year, or a history of myocardial infarction within the last 6 months prior to enrollment.
* Subject has neoplastic disease requiring therapy within 12 months prior to enrollment.
* Presence of clinically relevant hepatic dysfunction.
* Presence of clinically relevant renal dysfunction.
* Evidence of clinically relevant cardiovascular disorders.
* Subject has a QTcB interval of ³500msec at Screening or Baseline (Visit 1 or 2; repeated measurements within 1 hour).
* Subject has a history of chronic alcohol or drug abuse within the last 6 months.
* Subject has clinically significant laboratory results that, in the opinion of the investigator, would make the subject unsuitable for entry into the trial.
* Subject is pregnant or nursing, or is of child bearing potential but (i) not surgically sterile, or, (ii) not using adequate birth control methods (including at least one barrier method) or, (iii) not sexually abstinent, or (iv) subject is not at least two years post menopausal.
* Subject has any medical or psychiatric condition that, in the opinion of the investigator, can jeopardize or would compromise the subject's ability to participate in this trial.
* Subject has a known hypersensitivity to any components of the trial medication stated in this protocol.
* Subject has a previous diagnosis of narcolepsy, sleep apnea syndrome, rapid eye movement (REM) behavior disorder, restless legs syndrome, or periodic limb movement disorder.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2004-12; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Motor performance; Sleep disorders; Clinical Global Impression; Patient Global Impression; Safety & Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, Monheim, Germany

REFERENCES:
- [Result] Giladi N, Fichtner A, Poewe W, Boroojerdi B. Rotigotine transdermal system for control of early morning motor impairment and sleep disturbances in patients with Parkinson's disease. J Neural Transm (Vienna). 2010 Dec;117(12):1395-9. doi: 10.1007/s00702-010-0506-4. Epub 2010 Nov 16. PMID 21080009